CLINICAL TRIAL: NCT01953601
Title: A Phase III, Randomized, Placebo-Controlled, Parallel-Group, Double-Blind Clinical Trial to Study the Efficacy and Safety of MK-8931 (SCH 900931) in Subjects With Amnestic Mild Cognitive Impairment Due to Alzheimer's Disease (Prodromal AD)
Brief Title: Efficacy and Safety Trial of Verubecestat (MK-8931) in Participants With Prodromal Alzheimer's Disease (MK-8931-019)
Acronym: APECS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8931-019; 2012-005542-38 (EudraCT Number); 142502 (Registry Identifier: JAPIC-CTI); MK-8931-019 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-09-25; First posted 2013-10-01 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Amnestic Mild Cognitive Impairment; Alzheimer's Disease; Prodromal Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — verubecestat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) (Experimental): [Part 1] Verubecestat 12 mg once daily for 104 weeks in Part 1 (Base Study). [Part 2] Participants completing Part 1 and continuing to Part 2 (Extension Study) receive Verubecestat 12 mg once daily for an additional 260 weeks.
  Interventions: Drug: Verubecestat 12 mg (Parts 1 and 2)
- Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) (Experimental): [Part 1] Verubecestat 40 mg once daily for 104 weeks in Part 1 (Base Study). [Part 2] Participants completing Part 1 and continuing to Part 2 (Extension Study) receive Verubecestat 40 mg once daily for an additional 260 weeks.
  Interventions: Drug: Verubecestat 40 mg (Parts 1 and 2)
- Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2) (Placebo Comparator): [Part 1] Placebo once daily for 104 weeks in Part 1 (Base Study). [Part 2] Participants completing Part 1 and continuing to Part 2 (Extension Study) receive Verubecestat 40 mg once daily for an additional 260 weeks.
  Interventions: Drug: Verubecestat 40 mg (Parts 1 and 2); Other: Placebo (Part 1)

INTERVENTIONS:
Drug: Verubecestat 12 mg (Parts 1 and 2) — Verubecestat 12 mg oral tablet, given once daily.
  Other Names: MK-8931
  Arms: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2)
Drug: Verubecestat 40 mg (Parts 1 and 2) — Verubecestat 40 mg oral tablet, given once daily. Verubecestat 40 mg given to participants in Arm C continuing to study Part 2.
  Other Names: MK-8931
  Arms: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2); Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Other: Placebo (Part 1) — Placebo matching verubecestat, given once daily as an oral tablet.
  Arms: Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)

SUMMARY:
This study consists of two parts, Part 1 and Part 2. Part 1 assesses the efficacy and safety of verubecestat (MK-8931) compared with placebo administered for 104 weeks in the treatment of amnestic mild cognitive impairment (aMCI) due to Alzheimer's Disease (AD), also known as prodromal AD. Participants are randomized to receive placebo, or 12 mg or 40 mg verubecestat, once daily. The primary study hypothesis for Part 1 is that ≥1 verubecestat dose is superior to placebo with respect to the change from baseline in the Clinical Dementia Rating scale-Sum of Boxes (CDR-SB) score at 104 weeks. Participants completing Part 1 may choose to participate in Part 2, which is a long term double-blind extension to assess efficacy and safety of verubecestat administered for up to an additional 260 weeks. In Part 2, all participants receive either 12 mg or 40 mg verubecestat, once daily.

DETAILED DESCRIPTION:
As a result of protocol amendment, Study Part 2 will contain a Positron Emission Tomography (PET) imaging substudy to assess regional neurofibrillary tangle (NFT) expression.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of prodromal AD, including the following:

   1. History of subjective memory decline with gradual onset and slow progression for at least one year corroborated by an informant,
   2. Objective impairment in episodic memory by memory test performed at Screening,
   3. Does not meet criteria for dementia, AND
   4. Positive Screening amyloid imaging PET scan using [18F]flutametamol tracer or positive Screening CSF tau:amyloid-β42 (Aβ42) ratio (Participants with a prior positive amyloid imaging PET scan or a Screening PET scan with florbetaben or florbetapir may be enrolled without a Screening flutemetamol scan with Sponsor approval)
2. Able to read at a 6th grade level or equivalent
3. If participant is receiving an acetylcholinesterase inhibitor or memantine, the dose must have been stable for at least three months before Screening
4. Must have a reliable and competent trial partner/informant who has a close relationship with the participant and is willing to accompany the participant to all required trial visits, and to monitor compliance of the administration of the trial medication

Inclusion Criteria for Extension Period (Part 2):

1. Tolerated study drug and completed the initial 104-week period of the trial (Part 1)
2. Participant must have a reliable and competent trial partner who must have a close relationship with the subject

Exclusion Criteria:

1. History of stroke
2. Evidence of a clinically relevant neurological disorder other than the disease being studied (i.e., prodromal AD)
3. History of seizures or epilepsy within the last 5 years
4. Evidence of a clinically relevant or unstable psychiatric disorder, excluding major depression in remission
5. Participant is at imminent risk of self-harm or of harm to others
6. History of alcoholism or drug dependency/abuse within the last 5 years before Screening
7. Participant does not have a magnetic resonance imaging (MRI) scan obtained within 12 months of Screening and is unwilling or not eligible to undergo an MRI scan at the Screening Visit. With Sponsor approval, a head computed tomography (CT) scan may be substituted for MRI scan to evaluate eligibility
8. History of hepatitis or liver disease that has been active within the 6 months prior to Screening
9. Recent or ongoing, uncontrolled, clinically significant medical condition within 3 months of Screening
10. History of malignancy occurring within the 5 years before Screening, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or localized prostate carcinoma
11. Clinically significant vitamin B12 or folate deficiency in the 6 months before Screening
12. Use of any investigational drugs or participation in clinical trials within the 30 days before Screening
13. History of a hypersensitivity reaction to more than three drugs
14. Has human immunodeficiency virus (HIV) by medical history
15. Participant is unwilling or has a contraindication to undergo PET scanning including but not limited to claustrophobia, excessive weight or girth
16. History or current evidence of long QT syndrome, corrected QT (QTc) interval ≥470 milliseconds (for male participants) or ≥480 milliseconds (for female participants), or torsades de pointes
17. Close family member (including the trial partner, spouse or children) who is among the personnel of the investigational or sponsor staff directly involved with this trial

Exclusion Criteria for Extension Period (Part 2):

1. Participant is at imminent risk of self-harm or of harm to others
2. Has developed a recent or ongoing, uncontrolled, clinically significant medical or psychiatric condition
3. Results of safety assessments (e.g., laboratory tests) performed in participant at end of Part 1 that are clinically unacceptable to the Investigator
4. Has developed a form of dementia that is not AD
5. Has progressed to dementia due to AD per investigator diagnosis in the initial 104-week study (Part 1).

Exclusion Criteria for NFT PET Substudy (Part 2):

1. Had one or two PET scans with MK-6240 in the initial 104-week study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1454 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Voss T, Kost J, Mercer SP, Furtek C, Randolph C, Lines C, Egan MF, Cummings JL. Progression from Prodromal Alzheimer's Disease to Mild Alzheimer's Disease Dementia in the Verubecestat APECS Study: Adjudicating Diagnostic Transitions. J Alzheimers Dis. 2023;92(1):341-348. doi: 10.3233/JAD-220836. PMID 36744336
- [Derived] Dockendorf MF, Jaworowicz D, Humphrey R, Anderson M, Breidinger S, Ma L, Taylor T, Dupre N, Jones C, Furtek C, Kantesaria B, Bateman KP, Woolf E, Egan MF, Stone JA. A Model-Based Approach to Bridging Plasma and Dried Blood Spot Concentration Data for Phase 3 Verubecestat Trials. AAPS J. 2022 Apr 6;24(3):53. doi: 10.1208/s12248-022-00682-5. PMID 35384522
- [Derived] Wessels AM, Lines C, Stern RA, Kost J, Voss T, Mozley LH, Furtek C, Mukai Y, Aisen PS, Cummings JL, Tariot PN, Vellas B, Dupre N, Randolph C, Michelson D, Andersen SW, Shering C, Sims JR, Egan MF. Cognitive outcomes in trials of two BACE inhibitors in Alzheimer's disease. Alzheimers Dement. 2020 Nov;16(11):1483-1492. doi: 10.1002/alz.12164. Epub 2020 Oct 13. PMID 33049114
- [Derived] Egan MF, Kost J, Voss T, Mukai Y, Aisen PS, Cummings JL, Tariot PN, Vellas B, van Dyck CH, Boada M, Zhang Y, Li W, Furtek C, Mahoney E, Harper Mozley L, Mo Y, Sur C, Michelson D. Randomized Trial of Verubecestat for Prodromal Alzheimer's Disease. N Engl J Med. 2019 Apr 11;380(15):1408-1420. doi: 10.1056/NEJMoa1812840. PMID 30970186
- [Derived] Kennedy ME, Stamford AW, Chen X, Cox K, Cumming JN, Dockendorf MF, Egan M, Ereshefsky L, Hodgson RA, Hyde LA, Jhee S, Kleijn HJ, Kuvelkar R, Li W, Mattson BA, Mei H, Palcza J, Scott JD, Tanen M, Troyer MD, Tseng JL, Stone JA, Parker EM, Forman MS. The BACE1 inhibitor verubecestat (MK-8931) reduces CNS beta-amyloid in animal models and in Alzheimer's disease patients. Sci Transl Med. 2016 Nov 2;8(363):363ra150. doi: 10.1126/scitranslmed.aad9704. PMID 27807285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N=1454 participants with prodromal Alzheimer's Disease (AD) were randomized, with N=1451 receiving study treatment.
Pre-assignment Details: This trial was conducted in 2 parts: a Base Study (Part 1), followed by an Extension Study (Part 2). Participants completing Part 1 had the option to continue to Part 2.
Period: Part 1 (Base Study)
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Started | 485 | 484 | 485
Treated | 483 | 484 | 484
Completed | 234 | 231 | 239
Not Completed | 251 | 253 | 246
Not completed — Adverse Event | 24 | 37 | 15
Not completed — Death | 2 | 0 | 3
Not completed — Lack of Efficacy | 3 | 1 | 4
Not completed — Lost to Follow-up | 1 | 3 | 6
Not completed — Non-compliance with study drug | 0 | 3 | 1
Not completed — Physician Decision | 3 | 7 | 4
Not completed — Screen failure | 1 | 0 | 1
Not completed — Site discontinued study participation | 2 | 0 | 0
Not completed — Study terminated by sponsor | 174 | 169 | 179
Not completed — Discontinued due to caregiver withdrawal | 7 | 8 | 10
Not completed — Subject moved | 2 | 2 | 1
Not completed — Withdrawal by Subject | 32 | 23 | 22
Period: Part 2 (Extension Study)
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Started | 198 (Number started refers only to participants completing Part 1, volunteering to continue to Part 2.) | 191 (Number started refers only to participants completing Part 1, volunteering to continue to Part 2.) | 204 (Number started refers only to participants completing Part 1, volunteering to continue to Part 2.)
Treated | 197 | 191 | 204
Completed | 0 | 0 | 0
Not Completed | 198 | 191 | 204
Not completed — Adverse Event | 1 | 1 | 10
Not completed — Death | 0 | 3 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 2
Not completed — Site discontinued study participation | 0 | 1 | 1
Not completed — Study terminated by sponsor | 185 | 178 | 187
Not completed — Discontinued due to caregiver withdrawal | 1 | 3 | 0
Not completed — Subject moved | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2) | Total
Number analyzed (Participants) | 485 | 484 | 485 | 1454
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.7 (7.1) | 71.0 (7.4) | 71.6 (7.1) | 71.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 244 | 213 | 686
  Male | 256 | 240 | 272 | 768
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 29 | 29 | 86
  Not Hispanic or Latino | 441 | 439 | 441 | 1321
  Unknown or Not Reported | 16 | 16 | 15 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 79 | 85 | 84 | 248
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 6 | 14
  White | 397 | 392 | 391 | 1180
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 2 | 3 | 2 | 7
Geographic Region [Count of Participants; unit: Participants] — Population: Includes all randomized participants receiving ≥1 dose of study treatment.
  Participants
    number analyzed (Participants) | 483 | 484 | 484 | 1451
    United States / Canada | 226 | 224 | 226 | 676
    Japan | 57 | 60 | 59 | 176
    Europe / Australia / New Zealand | 163 | 163 | 161 | 487
    Other | 37 | 37 | 38 | 112
APOE4 Genotype [Count of Participants; unit: Participants] — Apolipoprotein E (APOE) genotype is the strongest genetic predictor of risk for developing AD. The number of participants testing positive or negative for the APOE4 allele at baseline is presented. Population: Includes all randomized participants receiving ≥1 dose of study treatment.
  Participants
    number analyzed (Participants) | 483 | 484 | 484 | 1451
    Negative | 155 | 146 | 148 | 449
    Positive | 328 | 337 | 335 | 1000
    Missing | 0 | 1 | 1 | 2
Baseline Use of Vitamin E [Count of Participants; unit: Participants] — The number of participants receiving Vitamin E (> or ≤ 400 International Units [IU] / day; or no use) is presented. Population: Includes all randomized participants receiving ≥1 dose of study treatment.
  Participants
    number analyzed (Participants) | 483 | 484 | 484 | 1451
    No Use | 351 | 372 | 355 | 1078
    ≤400 IU / day | 123 | 100 | 120 | 343
    >400 IU / day | 9 | 12 | 9 | 30
Background Alzheimer's Disease (AD) Treatment [Count of Participants; unit: Participants] — The number of participants receiving acetylcholinesterase inhibitors (AChEI) and/or memantine (or no background AD treatment) is presented. Population: Includes all randomized participants receiving ≥1 dose of study treatment.
  Participants
    number analyzed (Participants) | 483 | 484 | 484 | 1451
    Use of AChEI alone | 182 | 191 | 180 | 553
    Use of memantine alone | 9 | 8 | 8 | 25
    Use of AChEI and memantine | 31 | 26 | 34 | 91
    No use of AChEI or memantine | 261 | 259 | 262 | 782
Mini-Mental State Examination (MMSE) Score [Count of Participants; unit: Participants] — The MMSE is a cognitive assessment of 5 domains (orientation; attention; memory; language; constructional praxis), with 11 questions scored based on number of correct responses. Depending on the question, scores range from 0 (no correct response) to either 1 (4 questions), 2 (1 question), 3 (3 questions), or 5 (3 questions). Scores for each question sum to a total MMSE score (range: 0-30); lower scores indicate worse cognitive performance. Participants are stratified by MMSE score (≥24-26 or ≥27) to ensure a representative population by AD severity across study arms. Population: Includes all randomized participants receiving ≥1 dose of study treatment.
  Participants
    number analyzed (Participants) | 483 | 484 | 484 | 1451
    MMSE ≥27 | 212 | 211 | 214 | 637
    MMSE ≥24-26 | 270 | 271 | 270 | 811
    Missing | 1 | 2 | 0 | 3
Clinical Dementia Rating Sum of Boxes (CDR-SB) Score [Mean (Standard Deviation); unit: Score on a Scale] — The CDR-SB score is a clinical rating of global cognitive function, comprised of 6 domains: memory; orientation; judgment and problem solving; community affairs; home and hobbies; and personal care. For each domain, the degree of impairment is assessed by a semi-structured interview of the participant as well as the participant's caregiver. For each domain, potential scores range from 0 (no impairment) to 3 (severe impairment). Individual domain scores are summed to a total CDR-SB score (range: 0-18). Higher scores indicate more severe cognitive impairment. Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose CDR-SB observation; and 2) tested positive for cortical amyloid load by positron emission tomography (PET).
  Score on a Scale
    number analyzed (Participants) | 465 | 458 | 469 | 1392
    (all) | 2.7 (1.3) | 2.7 (1.3) | 2.6 (1.2) | 2.66 (1.25)
Composite Cognition Score-3 Domain (CCS-3D) [Mean (Standard Deviation); unit: Z-score] — CCS-3D is composed of individual cognitive tests, grouped into 3 domains: 1) episodic memory; 2) executive function; and 3) attention/processing speed. For each cognitive test, a z-score (Z) is calculated at each time point [Z = (observed value - study population mean at baseline) / study population standard deviation at baseline]. These individual Zs are first combined into domain-specific Zs, and then into a composite Z, (i.e. CCS-3D). Theoretically, 99.9% of CCS-3D will be ± 3; more positive CCS-3D indicate greater cognitive impairment relative to the total study population at baseline. Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose CCS-3D observation; and 2) tested positive for cortical amyloid load by PET.
  Z-score
    number analyzed (Participants) | 441 | 424 | 440 | 1305
    (all) | 0.0 (1.0) | 0.0 (1.0) | -0.1 (1.0) | -0.01 (1.00)
Total Hippocampal Volume (THV) [Mean (Standard Deviation); unit: µL] — THV was measured by volumetric magnetic resonance imaging (vMRI). Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose THV observation; and 2) tested positive for cortical amyloid load by PET.
  µL
    number analyzed (Participants) | 168 | 181 | 191 | 540
    (all) | 6448.4 (1107.1) | 6468.5 (1105.8) | 6435.4 (987.2) | 6450.55 (1063.87)
[18F]Flutemetamol Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVR) [Mean (Standard Deviation); unit: Standard Uptake Value Ratio (SUVR)] — [18F]Flutemetamol PET SUVR measures brain cortical amyloid load. The PET tracer [18F]Flutemetamol was given intravenously (IV). After 90 minutes uptake, participants were scanned for 20 minutes. Using the PET scan images, SUVRs, the ratio of tracer signal in a specific region compared to a reference region (RR; subcortical white matter) are calculated for brain regions of interest (ROIs). SUVRs from a selected set of brain regions are averaged to compute a composite SUVR. Higher composite SUVR values indicate increased amyloid load in selected brain regions. Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose SUVR observation; and 2) tested positive for cortical amyloid load by PET. SUVR testing occurred at select sites as a Part 1 substudy.
  Standard Uptake Value Ratio (SUVR)
    number analyzed (Participants) | 63 | 59 | 65 | 187
    (all) | 0.86 (0.07) | 0.87 (0.07) | 0.85 (0.06) | 0.86 (0.07)
AD Cooperative Study-Activities of Daily Living, Mild Cognitive Impairment (ADCS-ADL MCI) Score [Mean (Standard Deviation); unit: Score on a Scale] — The ADCS-ADL MCI is an 18-item assessment of recent, observed performance of activities of daily living administered to participants' trial partners in an interview format. For the 18 items, scores range from 0 (no independence) to (depending on the item) either 2 (5 items), 3 (9 items), or 4 (4 items), with higher scores indicating greater independence in activity performance. Scores from individual items are summed for a total ADCS-ADL score (range: 0-53). Lower scores indicate less independence in activity performance and, as a result, greater AD severity. Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose ADCS-ADL MCI observation; and 2) tested positive for cortical amyloid load by PET.
  Score on a Scale
    number analyzed (Participants) | 469 | 462 | 472 | 1403
    (all) | 42.2 (5.9) | 43.1 (5.4) | 42.8 (5.9) | 42.71 (5.73)
Cerebrospinal Fluid (CSF) Total Tau Concentration [Mean (Standard Deviation); unit: pg/mL] — Total Tau concentration in the CSF was monitored as a measure of brain tau pathology. Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose observation for CSF Total Tau concentration; and 2) tested positive for cortical amyloid load by PET. CSF Total Tau concentration was analyzed at select trial sites as a Part 1 substudy.
  pg/mL
    number analyzed (Participants) | 5 | 6 | 6 | 17
    (all) | 203.8 (129.1) | 159.3 (79.0) | 243.5 (97.0) | 202.12 (101.91)

OUTCOME MEASURES:

1. Primary Outcome: Part 1 (Base Study). Least Squares Mean (LSM) Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) Score at Week 104
Description: LSM change from baseline at week 104 was assessed for CDR-SB score, a clinical rating of global cognitive function, comprised of 6 domains: memory; orientation; judgment and problem solving; community affairs; home and hobbies; and personal care. For each domain, the degree of impairment is assessed by a semi-structured interview of the participant as well as the participant's caregiver. For each domain, potential scores range from 0 (no impairment) to 3 (severe impairment). Individual domain scores are summed to a total CDR-SB score (range: 0-18). Higher scores indicate more severe cognitive impairment. Further, increases in cognitive impairment would be reflected by increases in CDR-SB score.
Time Frame: Baseline and Week 104 in Part 1
Population: Includes all participants receiving ≥1 dose of study treatment in Part 1 who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose CDR-SB observation; and 2) tested positive for cortical amyloid load by PET.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 465 | 458 | 469
Score on a Scale | 1.6 [1.4 to 1.9] | 2.0 [1.8 to 2.3] | 1.6 [1.3 to 1.8]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.6734, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = 0.1, 97.51% CI 2-sided [-0.3 to 0.4] — Difference in LSM = Arm A - Arm C; Analysis model includes categorical factors of geographic region, time, treatment, gender, APOE genotype, baseline use of Vitamin E, baseline use of AChEI, and the interaction of time by treatment, with baseline value, the interaction of baseline value and time, the baseline value of MMSE and the baseline value of age included as continuous covariates
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.0141, Longitudinal ANCOVA; Difference in Least Squares Means (LSM) = 0.4, 97.51% CI 2-sided [0.0 to 0.8] — Difference in LSM = Arm B - Arm C; [other analysis details as in outcome 1, analysis 1]

2. Primary Outcome: Part 2 (Extension Study). Mean Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) Score at Week 130
Description: Mean change from baseline at week 130 was assessed for CDR-SB score, a clinical rating of global cognitive function, comprised of 6 domains: memory; orientation; judgment and problem solving; community affairs; home and hobbies; and personal care. For each domain, the degree of impairment is assessed by a semi-structured interview of the participant as well as the participant's caregiver. For each domain, potential scores range from 0 (no impairment) to 3 (severe impairment). Individual domain scores are summed to a total CDR-SB score (range: 0-18). Higher scores indicate more severe cognitive impairment. Further, increases in cognitive impairment would be reflected by increases in CDR-SB score. Per protocol, baseline refers to the baseline measurement obtained in Part 1.
Time Frame: Baseline and Week 130 (i.e., Week 26 of Part 2)
Population: All randomized participants continuing to Part 2, with: 1) both a pre-dose baseline and ≥1 within-analysis-window, post-dose CDR-SB observation; 2) a positive test for cortical amyloid load by PET; and 3) a CDR-SB observation at week 130.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 120 | 113 | 124
Score on a Scale | 2.0 (2.5) | 1.9 (2.2) | 1.5 (2.1)

3. Primary Outcome: Part 1 (Base Study). Percentage of Participants Who Experienced ≥1 Adverse Event (AE)
Description: The percentage of participants experiencing an AE in Part 1 was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: Up to Week 106 (up to 2 weeks following cessation of study treatment in Part 1)
Population: All randomized participants in Part 1, receiving ≥1 dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 483 | 484 | 484
Percentage of Participants | 91.3 | 92.1 | 87.0
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = 4.32, 95% CI 2-sided [0.40 to 8.31] — Difference in % = Arm A - Arm C
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = 5.17, 95% CI 2-sided [1.33 to 9.09] — Difference in % = Arm B - Arm C

4. Primary Outcome: Part 1 (Base Study). Percentage of Participants Who Discontinued From Study Drug Due to an Adverse Event (AE)
Description: The percentage of participants who discontinued from study drug due to an AE in Part 1 was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: Up to Week 104 in Part 1
Population: All randomized participants in Part 1, receiving ≥1 dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 483 | 484 | 484
Percentage of Participants | 6.6 | 10.1 | 4.5
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = 2.08, 95% CI 2-sided [-0.84 to 5.10] — Difference in % = Arm A - Arm C
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = 5.58, 95% CI 2-sided [2.35 to 8.99] — Difference in % = Arm B - Arm C

5. Primary Outcome: Part 2 (Extension Study). Percentage of Participants Who Experienced ≥1 Adverse Event (AE)
Description: The percentage of participants experiencing an AE in Part 2 was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: From Week 104 (start of treatment in Part 2) up to Week 210 (up to 2 weeks following cessation of study treatment in Part 2)
Population: All randomized participants continuing to Part 2, receiving ≥1 dose of trial treatment in Part 2. For included participants, the data reflect AEs occurring in Part 2 only.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 197 | 191 | 204
Percentage of Participants | 59.4 | 55.5 | 66.2
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = -6.79, 95% CI 2-sided [-16.16 to 2.68] — Difference in % = Arm A - Arm C
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = -10.68, 95% CI 2-sided [-20.16 to -1.04] — Difference in % = Arm B - Arm C

6. Primary Outcome: Part 2 (Extension Study). Percentage of Participants Who Discontinued From Study Drug Due to an Adverse Event (AE)
Description: The percentage of participants who discontinued from study drug due to an AE in Part 2 was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: From Week 104 (start of treatment in Part 2) up to Week 208 (i.e., up to Week 104 in Part 2)
Population: All randomized participants continuing to Part 2, receiving ≥1 dose of trial treatment in Part 2. For included participants, the data reflect discontinuations occurring in Part 2 only.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 197 | 191 | 204
Percentage of Participants | 1.0 | 1.0 | 3.4
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = -2.42, 95% CI 2-sided [-6.03 to 0.61] — Difference in % = Arm A - Arm C
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Other; Difference in % vs Placebo = -2.38, 95% CI 2-sided [-6.01 to 0.71] — Difference in % = Arm B - Arm C

7. Secondary Outcome: Part 1 (Base Study). Event-Rate Per 100 Participant Years for Progression to a Clinical Diagnosis of Probable AD Dementia
Description: The event-rate per 100 participant-years for progression to a clinical diagnosis of probable AD dementia was calculated. Adjudication of a potential case was triggered if either: 1) in the investigator's own expert judgment, they think the participant may have progressed to dementia and/or 2) the participant's CDR-SB score is ≥2 points higher compared to baseline. Cases of progression to probable AD dementia confirmed by an external adjudication committee were counted as events in the analysis. The event-rate was calculated as the number of events divided by total follow-up time (participant-years) x 100; unit of measure is event-rate / 100 participant-years.
Time Frame: Up to Week 104 in Part 1
Population: Includes all participants receiving ≥1 dose of study treatment in Part 1 who tested positive for cortical amyloid load by PET.
Measure: Number; unit: Event-Rate / 100 Participant-Years
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 480 | 481 | 481
Event-Rate / 100 Participant-Years | 24.5 | 25.5 | 19.3
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.0222, Regression, Cox; Hazard Ratio (HR) = 1.301, 97.51% CI 2-sided [1.005 to 1.684] — HR = Arm A / Arm C; Based on Cox regression model with Efron's method of tie handling with treatment, background AD treatment (use, no use), sex, APOE4 status (carrier, non-carrier) and baseline use of Vitamin E as categorical covariates and age and baseline MMSE value as continuous covariates
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.0050, Regression, Cox; Hazard Ratio (HR) = 1.382, 97.51% CI 2-sided [1.067 to 1.790] — HR = Arm B / Arm C; [other analysis details as in outcome 7, analysis 1]

8. Secondary Outcome: Part 1 (Base Study). Estimated Least Squares Mean Difference Between the Last (Week 104) and First (Week 13) Post-dose CDR-SB Assessment
Description: LSM difference between weeks 104 and 13 was estimated for CDR-SB score, a clinical rating of global cognitive function, comprised of 6 domains: memory; orientation; judgment / problem solving; community affairs; home / hobbies; and personal care. For each domain, degree of impairment is scored by a semi-structured interview of the participant and the participant's caregiver (domain score range: 0 [no impairment] to 3 [severe impairment]). Domain scores sum to a total CDR-SB score (range: 0-18); higher scores indicate more severe cognitive impairment. Further, increased cognitive impairment is reflected by higher CDR-SB scores; larger differences between week 104 and week 13 scores indicates accelerated AD progression.
Time Frame: Week 13 and Week 104 in Part 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 465 | 458 | 469
Score on a Scale | 1.5 [1.3 to 1.7] | 1.8 [1.5 to 2.0] | 1.5 [1.3 to 1.7]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.9109, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = 0.0, 97.51% CI 2-sided [-0.3 to 0.4] — Difference in LSM = Arm A - Arm C; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.0824, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = 0.3, 97.51% CI 2-sided [-0.1 to 0.7] — Difference in LSM = Arm B - Arm C; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: Part 1 (Base Study). Least Squares Mean Change From Baseline in the 3-Domain Composite Cognition Score (CCS-3D) at Week 104
Description: CCS-3D is composed of individual cognitive tests, grouped into 3 domains: 1) episodic memory; 2) executive function; and 3) attention/processing speed. For each cognitive test, a z-score (Z) is calculated at each time point [Z = (observed value - study population mean at baseline) / study population standard deviation at baseline]. These individual Zs are first combined into domain-specific Zs, and then into a composite Z, (i.e. CCS-3D). Theoretically, 99.9% of CCS-3D will be ± 3; more positive CCS-3D indicate greater cognitive impairment relative to the total study population at baseline. Further, negative changes in CCS-3D over time indicate improved cognition relative to the total study population at baseline.
Time Frame: Baseline and Week 104 in Part 1
Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose CCS-3D observation; and 2) tested positive for cortical amyloid load by PET.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 441 | 424 | 440
Z-score | 0.8 [0.7 to 0.9] | 0.8 [0.7 to 0.9] | 0.8 [0.7 to 0.9]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.9510, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = 0.0, 97.51% CI 2-sided [-0.2 to 0.2] — Difference in LSM = Arm A - Arm C; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.9392, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = 0.0, 97.51% CI 2-sided [-0.2 to 0.2] — Difference in LSM = Arm B - Arm C; [other analysis details as in outcome 1, analysis 1]

10. Secondary Outcome: Part 1 (Base Study). Least Squares Mean Percent Change From Baseline in Total Hippocampal Volume (THV) at Week 104
Description: Least squares mean percent change from baseline at week 104 was calculated for THV as measured by volumetric magnetic resonance imaging (vMRI). Negative percent changes from baseline indicate decreases in THV (i.e. increased hippocampal atrophy).
Time Frame: Baseline and Week 104 in Part 1
Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose THV observation; and 2) tested positive for cortical amyloid load by PET.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 168 | 181 | 191
Percent Change | -6.5 [-6.9 to -6.2] | -6.7 [-7.1 to -6.3] | -6.1 [-6.5 to -5.7]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.1133, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = -0.4, 97.51% CI 2-sided [-1.0 to 0.2] — Difference in LSM = Arm A - Arm C; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.0310, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = -0.6, 97.51% CI 2-sided [-1.2 to 0.0] — Difference in LSM = Arm B - Arm C; [other analysis details as in outcome 1, analysis 1]

11. Secondary Outcome: Part 1 (Base Study). Least Squares Mean Change From Baseline in Composite Cortical Amyloid Standard Uptake Value Ratio (SUVR) Assessed With Amyloid Tracer [18F]Flutemetamol Using Positron Emission Tomography (PET) Imaging at Week 104
Description: [18F]Flutemetamol PET SUVR measures brain cortical amyloid load. The PET tracer [18F]Flutemetamol was given intravenously (IV). After 90 minutes, participants were scanned for 20 minutes. Using the PET scan images, SUVRs, the ratio of tracer signal in a specific region compared to a reference region (RR; subcortical white matter) are calculated for brain regions of interest (ROIs). SUVRs from a selected set of brain regions are averaged to compute a composite SUVR. Higher composite SUVR values indicate increased amyloid load in selected brain regions, with negative changes in composite cortical SUVR over time indicating decreases in brain amyloid load.
Time Frame: Baseline and Week 104 in Part 1
Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose SUVR observation; and 2) tested positive for cortical amyloid load by PET.
Measure: Least Squares Mean (95% Confidence Interval); unit: Standard Uptake Value Ratio (SUVR)
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 63 | 59 | 65
Standard Uptake Value Ratio (SUVR) | -0.03 [-0.04 to -0.03] | -0.04 [-0.05 to -0.04] | 0.02 [0.02 to 0.03]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p < 0.0001, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = -0.05, 97.51% CI 2-sided [-0.06 to -0.04] — Difference in LSM = Arm A - Arm C; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p < 0.0001, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = -0.06, 97.51% CI 2-sided [-0.07 to -0.05] — Difference in LSM = Arm B - Arm C; [other analysis details as in outcome 1, analysis 1]

12. Secondary Outcome: Part 1 (Base Study). Least Squares Mean Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment Version) (ADCS-ADL MCI) Score at Week 104
Description: Least squares mean change from baseline at week 104 was assessed for the ADCS-ADL MCI score. The ADCS-ADL MCI is an 18-item assessment of recent, observed performance of activities of daily living administered to participants' trial partners in an interview format. For the 18 items, scores range from 0 (no independence) to (depending on the item) either 2 (5 items), 3 (9 items), or 4 (4 items), with higher scores indicating greater independence in activity performance. Scores from individual items sum to a total ADCS-ADL score (range: 0-53). Lower scores indicate less independence in activity performance and, as a result, greater AD severity. Further, increases in AD severity over time would be reflected by decreases in ADCS-ADL score.
Time Frame: Baseline and Week 104 in Part 1
Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose ADCS-ADL MCI observation; and 2) tested positive for cortical amyloid load by PET.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 469 | 462 | 472
Score on a Scale | -5.2 [-6.1 to -4.3] | -5.8 [-6.8 to -4.8] | -4.1 [-5.0 to -3.3]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.0960, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = -1.0, 97.51% CI 2-sided [-2.4 to 0.4] — Difference in LSM = Arm A - Arm C; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) vs Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2); Test type: Superiority; p = 0.0110, Longitudinal ANCOVA; Difference in Least Squares Mean (LSM) = -1.7, 97.51% CI 2-sided [-3.2 to -0.2] — Difference in LSM = Arm B - Arm C; [other analysis details as in outcome 1, analysis 1]

13. Secondary Outcome: Part 1 (Base Study). Mean Percent Change From Baseline in Cerebrospinal Fluid (CSF) Total Tau Concentration at Week 104
Description: Mean percent change from baseline at week 104 was calculated for Total Tau concentration in CSF, a measure of brain tau pathology. Per protocol, CSF Total Tau concentration was analyzed as part of a substudy in Part 1, with testing occurring only at select trial sites.
Time Frame: Baseline and Week 104 in Part 1
Population: Includes all participants receiving ≥1 dose of study treatment who: 1) had both a pre-dose baseline and ≥1 within-analysis-window, post-dose observation for CSF Total Tau concentration; and 2) tested positive for cortical amyloid load by PET. CSF Total Tau concentration was analyzed at select trial sites as a Part 1 substudy.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Arm A. Verubecestat 12 mg (Part 1); 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 1); 40 mg (Part 2) | Arm C. Placebo (Part 1); Verubecestat 40 mg (Part 2)
Number analyzed (Participants) | 5 | 6 | 6
Percent Change | 33.2 (44.3) | 42.8 (39.7) | 10.2 (27.9)

ADVERSE EVENTS:
Time Frame: [Part 1]: Up to Week 106 of Part 1 (up to 2 weeks following cessation of study treatment in Part 1); [Part 2]: From Week 104 (start of treatment in Part 2) up to Week 210 (up to 2 weeks following cessation of study treatment in Part 2).
Description: [Part 1] Includes all randomized participants in Part 1 (Base Study) receiving ≥1 dose of study treatment. [Part 2] Includes all randomized participants continuing to Part 2 (Extension Study) receiving ≥1 dose of study treatment in Part 2. For Part 2-specific arms, only the AEs occurring during Part 2 are reported.
Groups:
- Arm A. Verubecestat 12 mg (Part 1): [Part 1] Verubecestat 12 mg once daily for 104 weeks in Part 1 (Base Study).
- Arm B. Verubecestat 40 mg (Part 1): [Part 1] Verubecestat 40 mg once daily for 104 weeks in Part 1 (Base Study).
- Arm C. Placebo (Part 1): [Part 1] Placebo once daily for 104 weeks in Part 1 (Base Study).
- Arm A. Verubecestat 12 mg (Part 2): [Part 2] Participants completing Part 1 and continuing to Part 2 (Extension Study) receive verubecestat 12 mg once daily for an additional 260 weeks.
- Arm B. Verubecestat 40 mg (Part 2); Arm C. Verubecestat 40 mg (Part 2): [Part 2] Participants completing Part 1 and continuing to Part 2 (Extension Study) receive verubecestat 40 mg once daily for an additional 260 weeks.
Arm/Group | Arm A. Verubecestat 12 mg (Part 1) | Arm B. Verubecestat 40 mg (Part 1) | Arm C. Placebo (Part 1) | Arm A. Verubecestat 12 mg (Part 2) | Arm B. Verubecestat 40 mg (Part 2) | Arm C. Verubecestat 40 mg (Part 2)
All-Cause Mortality (participants affected / at risk) | 3/483 | 1/484 | 3/484 | 0/197 | 3/191 | 0/204
Serious Adverse Events (participants affected / at risk) | 124/483 | 101/484 | 96/484 | 10/197 | 22/191 | 24/204
Other Adverse Events (participants affected / at risk) | 221/483 | 223/484 | 202/484 | 39/197 | 31/191 | 40/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A. Verubecestat 12 mg (Part 1) (N=483) | Arm B. Verubecestat 40 mg (Part 1) (N=484) | Arm C. Placebo (Part 1) (N=484) | Arm A. Verubecestat 12 mg (Part 2) (N=197) | Arm B. Verubecestat 40 mg (Part 2) (N=191) | Arm C. Verubecestat 40 mg (Part 2) (N=204)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris aggravated (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation aggravated (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease aggravated (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Recurrent atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular bigeminy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign paroxysmal positional vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract bilateral NOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal upset (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids aggravated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Indirect inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left upper quadrant pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness epigastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain aggravated (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pressure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever of unknown origin (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacillus bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of foot (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of hand (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis of leg (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza B virus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prosthesis related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic arthritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bimalleolar fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruise of head (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Finger injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture of intertrochanteric section of femur, closed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured mandible (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Joint ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spine compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Olecranon fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain trauma activated (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid bleeding (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (traumatic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture T12 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trochanteric femoral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal occult blood (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia aggravated (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical spondylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herniated nucleus pulposus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hips osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis aggravated (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (14) | 8 (10) | 6 (7) | 4 (4) | 2 (2) | 3 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoma in situ of breast ductal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic tubular adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lentigo melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodular basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreas cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Prostate carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 3 (4) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Squamous cell carcinoma of skin well differentiated (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the nasal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urothelial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complex partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia aggravated (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epileptic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Felt faint (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurocardiogenic syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nonconvulsive status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncopal attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tremor aggravated (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion aggravated (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis aggravated (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic episode (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatisation disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unsuccessful suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus renal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stone urinary bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteral stricture (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urogenital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Collapse of lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exanthem (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticarial rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive episode (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral obliterative arteriopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticular disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyloric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza A virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurologic reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A. Verubecestat 12 mg (Part 1) (N=483) | Arm B. Verubecestat 40 mg (Part 1) (N=484) | Arm C. Placebo (Part 1) (N=484) | Arm A. Verubecestat 12 mg (Part 2) (N=197) | Arm B. Verubecestat 40 mg (Part 2) (N=191) | Arm C. Verubecestat 40 mg (Part 2) (N=204)
Diarrhoea (Gastrointestinal disorders) | 28 (35) | 21 (22) | 36 (38) | 6 (7) | 2 (2) | 3 (3)
Cold (Infections and infestations) | 16 (20) | 25 (28) | 24 (34) | 1 (1) | 4 (4) | 3 (3)
Common cold syndrome (Infections and infestations) | 22 (33) | 32 (48) | 26 (38) | 9 (10) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 31 (37) | 21 (24) | 31 (38) | 3 (4) | 6 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 30 (37) | 26 (35) | 23 (30) | 3 (3) | 3 (4) | 8 (10)
Fall (Injury, poisoning and procedural complications) | 42 (56) | 36 (48) | 33 (41) | 8 (8) | 6 (8) | 7 (10)
Weight decreased (Investigations) | 27 (27) | 32 (32) | 10 (10) | 6 (6) | 0 (0) | 8 (8)
Dizziness (Nervous system disorders) | 37 (49) | 31 (36) | 25 (25) | 4 (4) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 32 (36) | 26 (27) | 24 (28) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 17 (17) | 28 (29) | 13 (15) | 3 (3) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 31 (48) | 40 (50) | 25 (26) | 6 (6) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT01953601/Prot_SAP_000.pdf